CLINICAL TRIAL: NCT01313117
Title: Dose Finding and Tolerability Study of Alpha-lipoic Acid in Patients at Risk for Paclitaxel Induced Peripheral Neuropathy
Brief Title: Alpha-lipoic Acid in Patients at Risk for Paclitaxel Induced Neuropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jeffrey Allen, Assistant Professor in Ken and Ruth Davee Department of Neurology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NUALA-01
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Results first posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Peripheral Neuropathy
Keywords: chemotherapy; peripheral neuropathy; paclitaxel; breast cancer
MeSH Terms: conditions — Peripheral Nervous System Diseases; Breast Neoplasms | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alpha lipoic acid (Experimental): Oral administration three times daily (morning, mid-day, night)
  Interventions: Drug: Alpha lipoic acid

INTERVENTIONS:
Drug: Alpha lipoic acid — The baseline dose is 100 mg three times daily for four months. Dose escalation will occur until a maximum tolerated dose is found.
  Other Names: Thioctic Acid

SUMMARY:
This study is being done because peripheral neuropathy, a condition that interrupts sensation in your limbs, is a common side effect of paclitaxel. There is some evidence that alpha lipoic acid (ALA), an antioxidant compound, protects neurons after exposure to paclitaxel. The purpose of this study is to assess the safety and tolerability of ALA and to find the best dose of ALA in patients that receive chemotherapy.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of Breast cancer.
2. Breast cancer must meet the following criteria:

   * Early stage breast cancer (stages I, IIA) must be estrogen receptor (ER) positive AND low tumor grade (histopathologic grade 1 or 2)
   * Locally advanced breast cancer (LABC) (stages IIB, IIIA, IIB as defined by the Union for International Cancer Control and American Joint Committee on Cancer) must be ER positive, HER2 positive or HER2 negative, AND satisfy the following requirements: high endocrine responsiveness (defined as greater than 50% of tumor cells staining for hormone receptors), Grade 1 or 2 histological grade, less than 4 nodes positive, absence of extensive peritumoral vascular invasion, AND pathological tumor size less than 5 cm.
   * Inflammatory breast cancer (IBC) (stage IIIC)
   * Metastatic breast cancer (stage IV)
3. Must be receiving single agent paclitaxel in their prescribed chemotherapy regimen.
4. Age > 18 years. There is no upper age limit for participation in this study.
5. Required lab values: AST, ALT, creatinine
6. Women of childbearing potential and sexually active males must agree to use contraception while on study.
7. ECOG performance status 0,1,2
8. All patients must have given signed, informed consent.

Exclusion Criteria

1. Breast cancer meeting the following criteria:

   * Breast cancer stage 0
   * Early stage breast cancer (stages I, IIA) that is ER negative OR higher tumor grade (histopathologic grade greater than 2)
   * Stages I, II, and IIIA triple negative breast cancer (negative for estrogen receptors, progesterone receptors, and HER2)
   * LABC (stages IIB, IIIA, IIB) if they have low endocrine responsiveness (defined as less than 50% of tumor cells staining for hormone receptors), Grade 3 histological grade, 4 or more nodes positive, presence of extensive peritumoral vascular invasion, OR pathological tumor size greater than 5 cm
   * LABC (stages IIB, IIIA, IIB) that are ER negative
2. Evidence of pre-existing peripheral neuropathy as determined by baseline Michigan neuropathy screening instrument score > 2.
3. Previous chemotherapy treatment of any kind.
4. AST and ALT >2 times upper limit of normal; Creatinine > 2.0 mg/dL.
5. Current use of medications or substances known to be associated with peripheral neuropathy.
6. Use of ALA or other anti-oxidant supplements during the prior three months.
7. Diabetes mellitus or use of medications known to lower blood sugar.
8. Participation in any other experimental trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Allen, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medical Faculty Foundation, Chicago, Illinois, United States

REFERENCES:
- [Background] Siau C, Xiao W, Bennett GJ. Paclitaxel- and vincristine-evoked painful peripheral neuropathies: loss of epidermal innervation and activation of Langerhans cells. Exp Neurol. 2006 Oct;201(2):507-14. doi: 10.1016/j.expneurol.2006.05.007. Epub 2006 Jun 22. PMID 16797537
- [Background] McCarty MF, Barroso-Aranda J, Contreras F. The "rejuvenatory" impact of lipoic acid on mitochondrial function in aging rats may reflect induction and activation of PPAR-gamma coactivator-1alpha. Med Hypotheses. 2009 Jan;72(1):29-33. doi: 10.1016/j.mehy.2008.07.043. Epub 2008 Sep 11. PMID 18789599
- [Background] Melli G, Taiana M, Camozzi F, Triolo D, Podini P, Quattrini A, Taroni F, Lauria G. Alpha-lipoic acid prevents mitochondrial damage and neurotoxicity in experimental chemotherapy neuropathy. Exp Neurol. 2008 Dec;214(2):276-84. doi: 10.1016/j.expneurol.2008.08.013. Epub 2008 Sep 9. PMID 18809400
- [Background] Ziegler D, Ametov A, Barinov A, Dyck PJ, Gurieva I, Low PA, Munzel U, Yakhno N, Raz I, Novosadova M, Maus J, Samigullin R. Oral treatment with alpha-lipoic acid improves symptomatic diabetic polyneuropathy: the SYDNEY 2 trial. Diabetes Care. 2006 Nov;29(11):2365-70. doi: 10.2337/dc06-1216. PMID 17065669
- [Background] Cremer DR, Rabeler R, Roberts A, Lynch B. Safety evaluation of alpha-lipoic acid (ALA). Regul Toxicol Pharmacol. 2006 Oct;46(1):29-41. doi: 10.1016/j.yrtph.2006.06.004. Epub 2006 Aug 14. PMID 16904799
- [Background] Segermann J, Hotze A, Ulrich H, Rao GS. Effect of alpha-lipoic acid on the peripheral conversion of thyroxine to triiodothyronine and on serum lipid-, protein- and glucose levels. Arzneimittelforschung. 1991 Dec;41(12):1294-8. PMID 1815532
- [Background] GAL EM, RAZEVSKA DE. Studies on the in vivo metabolism of lipoic acid. 1. The fate of DL-lipoic acid-S35 in normal and thiamine-deficient rats. Arch Biochem Biophys. 1960 Aug;89:253-61. doi: 10.1016/0003-9861(60)90051-5. No abstract available. PMID 13825981
- [Background] Cremer DR, Rabeler R, Roberts A, Lynch B. Long-term safety of alpha-lipoic acid (ALA) consumption: A 2-year study. Regul Toxicol Pharmacol. 2006 Dec;46(3):193-201. doi: 10.1016/j.yrtph.2006.06.003. Epub 2006 Aug 8. PMID 16899332
- [Background] Ziegler D, Hanefeld M, Ruhnau KJ, Meissner HP, Lobisch M, Schutte K, Gries FA. Treatment of symptomatic diabetic peripheral neuropathy with the anti-oxidant alpha-lipoic acid. A 3-week multicentre randomized controlled trial (ALADIN Study). Diabetologia. 1995 Dec;38(12):1425-33. doi: 10.1007/BF00400603. PMID 8786016
- [Background] Reljanovic M, Reichel G, Rett K, Lobisch M, Schuette K, Moller W, Tritschler HJ, Mehnert H. Treatment of diabetic polyneuropathy with the antioxidant thioctic acid (alpha-lipoic acid): a two year multicenter randomized double-blind placebo-controlled trial (ALADIN II). Alpha Lipoic Acid in Diabetic Neuropathy. Free Radic Res. 1999 Sep;31(3):171-9. doi: 10.1080/10715769900300721. PMID 10499773
- [Background] Ziegler D, Hanefeld M, Ruhnau KJ, Hasche H, Lobisch M, Schutte K, Kerum G, Malessa R. Treatment of symptomatic diabetic polyneuropathy with the antioxidant alpha-lipoic acid: a 7-month multicenter randomized controlled trial (ALADIN III Study). ALADIN III Study Group. Alpha-Lipoic Acid in Diabetic Neuropathy. Diabetes Care. 1999 Aug;22(8):1296-301. doi: 10.2337/diacare.22.8.1296. PMID 10480774
- [Background] Ruhnau KJ, Meissner HP, Finn JR, Reljanovic M, Lobisch M, Schutte K, Nehrdich D, Tritschler HJ, Mehnert H, Ziegler D. Effects of 3-week oral treatment with the antioxidant thioctic acid (alpha-lipoic acid) in symptomatic diabetic polyneuropathy. Diabet Med. 1999 Dec;16(12):1040-3. doi: 10.1046/j.1464-5491.1999.00190.x. PMID 10656234
- [Background] Ametov AS, Barinov A, Dyck PJ, Hermann R, Kozlova N, Litchy WJ, Low PA, Nehrdich D, Novosadova M, O'Brien PC, Reljanovic M, Samigullin R, Schuette K, Strokov I, Tritschler HJ, Wessel K, Yakhno N, Ziegler D; SYDNEY Trial Study Group. The sensory symptoms of diabetic polyneuropathy are improved with alpha-lipoic acid: the SYDNEY trial. Diabetes Care. 2003 Mar;26(3):770-6. doi: 10.2337/diacare.26.3.770. PMID 12610036

RESULTS

PARTICIPANT FLOW:
Period: Cohort 1: Dose Level 1 (ALA 300mg Daily)
Arm/Group | Alpha Lipoic Acid
Started | 2
Completed | 2
Not Completed | 0
Period: Cohort 2: Dose Level 2 (ALA 600mg Daily)
Arm/Group | Alpha Lipoic Acid
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1
Period: Cohort 3: Dose Level 3 (ALA 400mg Daily)
Arm/Group | Alpha Lipoic Acid
Started | 2
Completed | 2
Not Completed | 0
Period: Cohort 4: Dose Level 4 (ALA 500mg Daily)
Arm/Group | Alpha Lipoic Acid
Started | 2
Completed | 2
Not Completed | 0
Period: Cohort 5: Dose Level 2 (ALA 600mg Daily)
Arm/Group | Alpha Lipoic Acid
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Alpha Lipoic Acid
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 56.7 [47 to 67]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Identification of the Optimal Dose of ALA Based on Acceptable Adverse Event(AE) Profile
Description: Based on acceptable adverse event (AE) profile and continual reassessment method dose escalation.
Time Frame: 4 months
Population: Although our dose finding analysis suggested a maximum tolerated dose of 500mg daily, it should be noted that we failed to fully complete the Continual Reassessment Method (CRM) dose finding portion of the study. As such, we can not make confident dose finding statements on the basis of this trial.
Measure: Number; unit: mg
Arm/Group | Alpha Lipoic Acid
Number analyzed (Participants) | 9
mg | 500

2. Secondary Outcome: Proportion of Patients Who Complete the Proposed Regimen of Daily ALA
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Alpha Lipoic Acid
Number analyzed (Participants) | 9
participants | 7

3. Secondary Outcome: Cumulative Rate of Adverse Events
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Alpha Lipoic Acid
Number analyzed (Participants) | 9
participants | 9

4. Secondary Outcome: Total Neuropathy Score (TNS)
Description: The Total Neuropathy score (TNS) is a validated score that combines signs, symptoms, and very limited nerve conduction studies (NCS). It was designed to assess peripheral nerve function and has been used as an endpoint in clinical trials of toxic neuropathy. The TNS is a composite scale with a range of values from 0 (normal) to 28 (severely affected). It includes data from 7 different categories. Patients are asked to assess the severity of sensory symptoms on a scale of 0 (no symptoms) to 4 (symptoms above knees or elbows, or functionally disabling). Next, 4 examination categories are assessed. These include pin sensation, vibration sensation, deep tendon reflexes, and strength. Signs are scored from 0 to 4 depending on severity. The nerve conduction portion of the scale consists of measurements of a motor (peroneal) and sensory (sural) nerve. Motor and sensory responses are graded on a scale of 0 to 4 depending on the severity of an abnormality.
Time Frame: 4 months
Population: Failure to reach the MTD precluded our ability to perform any meaningful analysis of the TNS.
Groups:
- Alpha Lipoic Acid: The study was designed to first explore the optimal ALA dose. The baseline dose was 100 mg three times daily for four months. Dose escalation was to occur until a maximum tolerated dose (MTD) was found. Once the MTD was established we were then to enroll additional patients at the MTD for efficacy analysis. The study failed to reach the MTD. Only small numbers of patients were enrolled. As such, we were unable to perform any meaningful efficacy (TNS) analysis.
Arm/Group | Alpha Lipoic Acid
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Alpha Lipoic Acid
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha Lipoic Acid (N=9)
Nausea (Gastrointestinal disorders) | 3 (3) — mild - probably related to study drug Moderate - possibly related to study drug Severe - possibly related to study drug
Rash (Skin and subcutaneous tissue disorders) | 3 (3) — Mild - not related to study drug Moderate - possibly related to study drug
Indigestion (Gastrointestinal disorders) | 1 (1) — Mild - probably related to study drug
Constipation (Gastrointestinal disorders) | 1 (1) — Moderate - possibly related to study drug
Pain (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The small number of enrolled patients precluded any meaningful ALA dose finding or neuropathy prevention efficacy statements. A formal statistical analysis of the data was not able to be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes